CLINICAL TRIAL: NCT07159399
Title: Impact of a Pharmacist-Led Education Program on Medication Adherence and Treatment Effectiveness of Direct Oral Anticoagulants in Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: A Pharmacist-Led Education Program to Improve Adherence to Direct Oral Anticoagulants in Patients With Atrial Fibrillation
Acronym: PharmAD-AF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Chi-Chuan Wang, Associate Professor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202404014RINC; NHRI-EX114-11409PI (Other Grant/Funding Number: National Health Research Institutes)
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education (Experimental): Patients in this arm will receive a comprehensive DOAC education from trained pharmacists.
  Interventions: Behavioral: Pharmacist-led patient education
- Usual care (Placebo Comparator): Patients in this arm will receive only usual care, without pharmacists providing additional DOAC education materials.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Pharmacist-led patient education — Trained pharnacists will provide information on: (1) the indication and the reason of DOAC prescription, (2) the name and the appearance of the DOAC agent, (3) the dose, frequency, time of administration, (4) the mechanism of action, (5) management of missed doses, (6) potential side effects and self-monitoring, and (7) perioperative management. An education leaflet about DOACs will also be provided to improve patients' understanding about the use of DOACs.
  Arms: Patient education
Other: Usual Care — Patients in the usual care group will receive only usual care, without pharmacists providing additional DOAC education materials.
  Arms: Usual care

SUMMARY:
Atrial fibrillation (irregular heartbeat) increases the risk of stroke, and patients are commonly treated with direct oral anticoagulants (DOACs). However, when patients do not take these medications regularly, the drugs may not work effectively, increasing health risks.

In this study, called PharmAD-AF, specially trained pharmacists will meet with patients who have atrial fibrillation and are prescribed DOACs. They will offer personalized education and support to help patients take their medications as directed.

Researchers will compare groups of patients who receive this pharmacist-led education versus those who receive usual care. The main goals are to assess whether pharmacist support improves how consistently patients take their DOACs and how well the treatment prevents strokes while avoiding the side effects of DOAC therapy.

If successful, the study will demonstrate how pharmacist-led education can help patients stick to their treatment plan and reduce serious health risks, offering a practical way to improve heart-related care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have a confirmed diagnosis of AF
* are expected to begin DOAC therapy for at least 3 months for stroke prevention

Exclusion Criteria:

* cannot understand DOAC-related education due to low literacy, language barriers, or cognitive impairment
* have been on DOAC therapy for more than 6 months
* using DOACs in off-label regimens
* are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Medication adherence will be measured at 3 months and 6 months after the baseline visit.
  Patients' adherence to DOACs will be assessed using the Adherence to Refills and Medications Scale (ARMS).
  The ARMS is a 12-item scale, including eight items on medication-taking adherence and four items on refill adherence. The total score ranges from 12 to 48, with higher scores indicating greater barriers to adherence.
  Unit of Measure: Score (points).

SECONDARY OUTCOMES:
Composite thromboembolic events | Composite thromboembolic events will be measured at 1 year and 2 years after the baseline visit
  Incidence of systemic thromboembolism, defined as occurrence of ischemic stroke (IS), transient ischemic attack (TIA), myocardial infarction (MI), coronary artery disease (CAD), peripheral artery disease (PAD), or venous thromboembolism (VTE).
  Unit of Measure: Percentage of participants (%)
Composite major bleeding events | Composite bleeding events will be measured at 1 year and 2 years after the baseline visit
  Incidence of major bleeding events, including intracranial hemorrhage (ICH), gastrointestinal bleeding (GIB), and other major bleeding requiring hospitalization.
  Unit of Measure: Percentage of participants (%)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT07159399/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT07159399/ICF_001.pdf